CLINICAL TRIAL: NCT03375333
Title: How Point-of-Care Ultrasound Affects the Diagnostic Process in General Practice. A Prospective Follow-up Study.
Brief Title: How Point-of-Care Ultrasound Affects the Diagnostic Process in General Practice.
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Camilla Aakjær Andersen, MD, Aalborg University
Other Study IDs: RUGPAalborg GULD projektet
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Ultrasound; Diagnostics; General Practice
Keywords: ultrasound; diagnostics; general practice; family medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 20GPs: 20 general practitioners, who use ultrasound in the examination of patients.

SUMMARY:
This study explores how Point of Care Ultrasound (POC-US) is used in general practice in Denmark and how it affects the diagnostic process and treatment of patients.

Twenty general practitioners (GPs) will register information each time they use POC-US during a one month period. The information will include indications and frequencies of the performed POC-US examinations, change in tentative diagnosis, plan, and treatment before and after the use of POC-US in relation to confidence in the tentative diagnosis, findings and quality of the POC-US examination.

This is an observational study without any intervention.

DETAILED DESCRIPTION:
This is a prospective, observational study aiming to describe: How general practitioners use POC-US in their daily practice, how POC-US influences the diagnostic process, and how POC-US affects the treatment of the patients.

The Use of POC-US will be explored through indication, frequency, time consumption, modification, and findings in order to describe:

* Which organs the GPs scan, when using POC-US?
* Which tentative diagnoses entail the use of POC-US?
* If GPs intend to rule-in/rule-out or explore, when using POC-US?
* How often the GPs use POC-US?
* How often are the GPs able to produce POC-US pictures of relevant structures?
* How much time POC-US adds to the consultation?
* How often a difference in what the GP intends to scan and what POC-US is actually used for occurs (modification of the performed POC-US)?
* How often POC-US leads to a specific finding?

The influences of the diagnostic process will be explored through change in the tentative diagnosis and change in the GP's confidence in the tentative diagnosis. The aim is to describe:

* If POC-US changes the patient's tentative diagnosis
* If POC-US increases the GP's confidence in the tentative diagnosis
* The relationship between the GP's expression of confidence and change in the number of tentative diagnoses
* The relationship between change from symptom diagnoses to disease diagnoses and the GP's expression of confidence in the tentative diagnosis
* The relationship between specific organs scanned and the GP's expression of confidence in the tentative diagnosis

The effects on the treatment of patients will be explored through changes in the plan or treatment for the patient. The aim is to describe:

* If POC-US changes the GP's plan for the patient
* If POC-US changes the treatment for the patient
* The relationship between findings and change in the plan or treatment for the patient.

Study setting:

The study will take place in 20 different general practices in Denmark where the GPs use POC-US.

Interventions

There is no intervention in this study since the GPs are already using POC-US in their examination of patients.

Sample size

There are around 75 GPs in Denmark, who use POC-US. Of those 20 GPs will be included in this study.

It is estimated that the GPs will use POC-US 2-3 times a day, and assuming a participation rate of 80%, there will be 640-960 US scan during the study period of one month.

Recruitment

Participating GPs:

GPs using POC-US will be recruited through the continuous medical educations small-groups program, US networks, conferences, through teaching sessions, and through contacts via the Danish general practice research units. Interested GPs will be asked to register and answer a questionnaire including background information concerning demography,education and use of ultrasound. The participating GPs will be selected randomly among these registrations after considering in-and exclusion criteria.

Participating patients:

Each time the participating GP use POC-US, he/she will ask the patient for informed consent. No restrictions are made regarding age or gender.

Base-line assessment of GPs

The GPs' technical skills will be evaluated at baseline using a standardized protocol (OSAUS).

Data collection

The registration tool will be developed as a questionnaire to be used before and after the GP uses POC-US in the consultation. The questionnaire will include a time log to ensure the before and after registration. Several pilot tests will be performed both in the research group and with GPs using POC-US in order to ensure comprehension, feasibility and compliance.

The GPs will be asked to access a questionnaire in the online database SurveyXact each time they use their ultrasound device during their daily work. The GPs can access the questionnaire on their mobile phone, iPad or computer, using a unique link (respondent link) allocated each participating GP. A key file, connecting each participating GP with the respondent link in Surveyxact (link), will be safely stored at the Research Unit for General Practice in Aalborg.

The GPs will give each patient a unique ID-number A Key file connecting this ID-number and the patients CPR-number (Danish national social security number) will be safely stored at the GP's clinic.

Before questions:

* GP ID number
* Patient ID number
* Date
* Patient gender
* Patient Age
* What is the main reason to use POC-US in this patient? (Rule-in/Rule-out or Explore)
* Which organs/positions is expected to be scanned? (organs on list)
* What is the main tentative diagnosis for this patient? (ICPC2 codes)
* Are there any other possible tentative diagnoses in this case? (ICPC2 codes)
* What is the overall plan for this patient? (Acute admission to hospital, Subacute referral to hospital, Elective referral hospital, Subacute referral to specialist, Elective referral to specialist, Referral to radiology, Other referral e.g. physiotherapist, Follow-up in the clinic, No plan for follow-up, Other)
* Which treatment will be initiated at this stage? (medical treatment, referral for treatment, initiated other treatment, None, Other)

After questions:

* time used on the POC-US examination? (minutes)
* Which organs/positions were scanned? (organs on list)
* Was the GP able to produce ultrasound images of the relevant structures of (inserted text) ? (yes, no - please specify)
* What did the GP find? (Certain positive findings, Uncertain positive findings, Certain negative findings, Uncertain negative findings, Incidental findings - please specify in free text)
* Before POC-US the following tentative diagnoses were registered (inserted text) Has this changed? (yes but the ICPC2 code is unchanged, Yes both diagnosis and ICPC2 code have changed, no)
* What is the tentative diagnosis for this patient now? (ICPC2 codes)
* Are there any other possible tentative diagnoses for this patient (please specify)? (ICPC2 codes)
* How is the GPs confidence in their main tentative diagnosis, after POC-US? (Highly increased confidence, More confident, unchanged confidence, Less confident, Highly reduced confidence)
* Before POC-US the following plan was registered (inserted text) for the patient. Has this plan changed? (yes, no)
* What is the overall plan for this patient, now? (Acute admission to hospital, Subacute referral to hospital, Elective referral hospital, Subacute referral to specialist, Elective referral to specialist, Referral to radiology, Other referral e.g. physiotherapist, Follow-up in the clinic, No plan for follow-up, Other)
* Before POC-US the following treatment was registered (inserted text) for the patient. Has the treatment changed? (yes, no)
* Which treatment will be initiated at this stage? (medical treatment, referral for treatment, initiated other treatment, None, Other)

Patient experience:

After the consultation, patients will be asked to complete a questionnaire about their experience with POC-US in the consultation. (This questionnaire will be described in detail in a separate protocol).

Follow-up

The GPs will be asked to save patient information on the included patients (Key file) in order to identify the patient for an additional follow-up after six months (described in a separate protocol).

Statistics

Descriptive statistics will be used. A prospective statistical analysis plan will be uploaded to clinical trials before datacollection begins.

Research ethics approval

The study is approved by the Danish Data Protection Agency and the Committee of Multipractice Studies in General Practice.

Since the study is an observational study and does not include any intervention, approval by the Danish National Committee on Health Research Ethics have been exempted.

Protocol amendments

Will be declared and all editions and changes of the protocol will be saved.

For further information a full protocol is uploaded to clinical trials.

ELIGIBILITY:
Inclusion Criteria (general practitioners):

1. Broad use of ultrasound
2. Working week of minimum four days
3. A minimum of 1400 patients listed
4. A minimum of two scanning probes
5. Previous participation in formal education in the use of ultrasound
6. Minimum six months experience with ultrasound in general practice.
7. Estimated use of ultrasound on a daily basis (average)

Exclusion Criteria (general practitioners):

1. Ultrasound device more than 10 years old
2. Conflict of interest, e.g. if the GP is part of the research group or if the GP has direct financial interest in selling US devices.
3. If less than five patients have been enrolled.

Inclusion/Exclusion criteria (patients):

All patients who consult the participating GP for conditions relevant for a POC-US examination will be offered to participate in the study. Patients are excluded if they do not wish to participate or if they are not able to give an informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participating GP practices will be selected purposively aiming at a difference in organisation, geography, and equipment. GPs will be selected to vary in experience both regarding seniority as GPs and experience of using POC-US. Thus we will include partnerships and solo practices, urban and rural practices as well as practices with variable number of probes and type of ultrasound scanner.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
How general practitioners use POC-US in their daily practice: | 2018
  The GP's indication for using POC-US will be described through the frequencies of the GP's intention to rule-in/ rule-out or explore when using POC-US and through frequencies of the tentative diagnoses that entail the use of POC-US.
  POC-US frequency is calculated as the number of consultations with POC-US (numerator) relative to all GP face-to-face consultations (denominator) during the study period. The frequency of each POC-US examination (numerator) will be compared to all types of POC-US scans (denominator).
  The GPs will measure the time used for the POC-US examination. By the before and after registration of the organs intended to scan and the organ actually scanned, the extent of modification of POC-US to include e.g. opportunistic screening, can be estimated.
  The findings in POC-US are measured through the categorical variables: Certain positive findings, uncertain positive findings, certain negative findings, uncertain negative findings, and incidental findings.

SECONDARY OUTCOMES:
How POC-US influences the diagnostic process | 2018
  The GPs are asked to declare the tentative diagnoses as one main tentative diagnosis and other possible diagnoses before the use of POC-US. After the use of POC-US the GPs will be shown their "Before-US" tentative diagnoses and asked if these diagnoses have changed. If the diagnoses have changed, they will be asked to specify this.
  The tentative diagnoses are registered as ICPC-2 codes in the questionnaire. The GPs are asked to register any change in their confidence in the tentative diagnoses after the use of POC-US by choosing one of the following variables on an ordinal scale: Increased confidence, more confident, unchanged confidence, less confident, reduced confidence.
  To test the reliability of the GPs' declaration of confidence, we will examine if an increased confidence is correlated to specific organs scanned (Q2.2), a reduction in the total number of diagnoses (Q1.3, Q1.4, Q2.6 and Q2.7), or a change from symptom diagnosis to disease diagnosis.
How POC-US affects the treatment of the patients: | 2018
  The GPs register their plan for the patient by choosing one or more of the following categorical variables before using POC-US: Acute admission to hospital, subacute referral to hospital, normal referral to hospital, subacute referral to specialist, normal referral to specialist, referral for radiology, other referral e.g. to physiotherapist, follow-up in the clinic, no plan for follow-up, other.
  After using POC-US the GP is shown the "before POC-US plan for the patient" and asked if this plan has changed. If the plan has changed, the GP is asked to specify.
  The GPs register their initiated treatment before POC-US by choosing one or more of the following categorical variables: Referral for treatment in the secondary sector, medication, other treatment, no treatment, other. After using POC-US the GP is shown the "before POC-US planned treatment for the patient" and asked if this planned treatment has changed. If the planned treatment has changed, the GP is asked to specify.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bach Jensen, Professor, GP, PhD, Study Chair — Aalborg University
Locations (1):
- Research unit for general practice in Aalborg,department of clinical medicine Aalborg university, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andersen CA, Brodersen JB, Mainz J, Thomsen JL, Graumann O, Lokkegaard T, Jensen MB. Does point-of-care ultrasound examination by the general practitioner lead to inappropriate care? A follow-up study. Scand J Prim Health Care. 2025 Sep;43(3):613-625. doi: 10.1080/02813432.2025.2487095. Epub 2025 Apr 10. PMID 40207775
- [Derived] Aakjaer Andersen C, Brodersen J, Davidsen AS, Graumann O, Jensen MBB. Use and impact of point-of-care ultrasonography in general practice: a prospective observational study. BMJ Open. 2020 Sep 17;10(9):e037664. doi: 10.1136/bmjopen-2020-037664. PMID 32948563

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03375333/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03375333/SAP_002.pdf